CLINICAL TRIAL: NCT04897711
Title: Perceptual Training for Improved Intelligibility of Dysarthric Speech
Brief Title: Perceptual Training to Improve Listeners' Ability to Understand Speech Produced by Individuals With Dysarthria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11110; R21DC018867 (NIH)
Record Dates: First submitted 2021-05-10; First posted 2021-05-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dysarthria; Intelligibility, Speech
Keywords: dysarthria; motor speech disorders; intelligibility; perceptual training
MeSH Terms: conditions — Dysarthria; Speech Intelligibility

STUDY DESIGN:
Intervention Model Description: 300 listeners will be recruited and enrolled. Each participant will be randomly assigned to receive perceptual training with one of 5 speakers with dysarthria, such that 30-50 listeners will be assigned to each speaker with dysarthria. All listener participants will receive the perceptual training intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Perceptual training with a speaker with dysarthria - Amyotrophic Lateral Sclerosis (ALS) (Experimental): To examine the effect of perceptual training with different speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases. Speech samples from a single speaker with dysarthria are utilized for all three phases. In this arm, listener participants were assigned to Speaker 1 (mixed flaccid-spastic dysarthria due to amyotrophic lateral sclerosis)
  Interventions: Behavioral: Perceptual Training
- Perceptual training with a speaker with dysarthria - Ataxic 1 (Experimental): To examine the effect of perceptual training with different speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases. Speech samples from a single speaker with dysarthria are utilized for all three phases. In this arm, listener participants were assigned to Speaker 2 (Ataxic dysarthria due to cerebellar degeneration)
  Interventions: Behavioral: Perceptual Training
- Perceptual training with a speaker with dysarthria - Parkinson's disease (PD) 1 (Experimental): To examine the effect of perceptual training with different speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases. Speech samples from a single speaker with dysarthria are utilized for all three phases. In this arm, listener participants were assigned to Speaker 3 (hypokinetic dysarthria due to Parkinson's disease)
  Interventions: Behavioral: Perceptual Training
- Perceptual training with a speaker with dysarthria - Ataxic 2 (Experimental): To examine the effect of perceptual training with different speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases. Speech samples from a single speaker with dysarthria are utilized for all three phases. In this arm, listener participants were assigned to Speaker 4 (Ataxic dysarthria due to cerebellar degeneration)
  Interventions: Behavioral: Perceptual Training
- Perceptual training with a speaker with dysarthria - Parkinson's disease (PD) 2 (Experimental): To examine the effect of perceptual training with different speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases. Speech samples from a single speaker with dysarthria are utilized for all three phases. In this arm, listener participants were assigned to Speaker 5 (hypokinetic dysarthria due to Parkinson's disease)
  Interventions: Behavioral: Perceptual Training

INTERVENTIONS:
Behavioral: Perceptual Training — Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
  Other Names: Familiarization

SUMMARY:
There exist very few effective treatments that ease the intelligibility burden of dysarthria. Perceptual training offers a promising avenue for improving intelligibility of dysarthric speech by offsetting the communicative burden from the speaker with dysarthria on to their primary communication partners-family, friends, and caregivers. This project, utilizing advanced explanatory models, will permit identification of speaker and listener parameters, and their interactions, that allow perceptual training paradigms to be optimized for intelligibility outcomes in dysarthria rehabilitation. This work addresses this critical gap in clinical practice and sets the stage for extension of dysarthria management to listener-targeted remediation-advancing clinical practice and enhanced communication and quality of life outcomes for this population.

DETAILED DESCRIPTION:
There exist very few effective treatments that ease the intelligibility burden of dysarthria, and all of these require cognitive and physical effort on the part of the speaker to achieve and maintain gains. Therefore, individuals with intelligibility deficits whose cognitive and physical impairments limit their ability to modify their speech are currently not viable treatment candidates. This constitutes a significant health disparity that disproportionately affects those clinical populations with developmental, cognitive, and/or significant neuromuscular impairment.

To address this critical gap in current dysarthria management, the weight of behavioral change is shifted from the speaker to the listener. While a novel concept for dysarthria management, the idea is firmly rooted in the field of psycholinguistics and supported by a programmatic body of research showing that listener-targeted perceptual training paradigms (wherein listeners are familiarized with the degraded speech signal and provided with an orthographic transcription of what the speaker is saying) result in statistically and clinically significant intelligibility gains in dysarthria. Further, preliminary evidence suggests that these intelligibility outcomes may be influenced by hypothesis-driven speaker parameters, such as acoustic predictability of speech rhythm cues, and listener parameters, such as expertise in rhythm perception.

A requisite next step to bringing listener-targeted perceptual training closer to clinical implementation, and the overarching goal of this clinical trial, is the systematic and rigorous analysis of the speaker and listener parameters, and their interactions, that modulate, and in some cases optimize, perceptual training benefits of intelligibility improvement. To achieve this aim, an existing database of dysarthric speech (20 speakers with dysarthria) and a large cohort of listeners (n = 400) across two well-established testing sites, Utah State University and Florida State University are utilized. Thus, the key deliverable resulting from this work will be explanatory models that account for the unique and joint contributions of speaker and listener parameters on the magnitude of intelligibility improvement following perceptual training with dysarthric speech.

ELIGIBILITY:
Inclusion Criteria:

*Native speakers of American English

Exclusion Criteria:

* No self-reported history of speech impairment
* No self-reported history of language impairment
* No self-reported history of cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Borrie, PhD, Principal Investigator — Utah State University; Kaitlin L Lansford, PhD, Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Utah State University, Logan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Results of the proposed research will be disseminated through conference presentations and manuscripts submitted to academic journals. In addition, the de-identified data will be available for public access via a data repository at the University of Michigan (ICPSR). The study will be registered in ClinicalTrials.gov within 21 days of enrollment of the first participant. Results will be submitted within 1 year of completion of the study. Informed consent documents will contain a statement concerning posting of information to ClinicalTrials.gov. Utah State University's Investigator Handbook (Chapter 9) outlines a policy for reporting all ClinicalTrials.gov information, specifically stating that it is the PI's responsibility to do so according to NIH policy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within one year of completion
Access Criteria: Information related to the protocol and statistical analysis plan will be shared in future publications. The analytic code will be shared via the Open Science website, with the link included in associated publications.

REFERENCES:
- [Background] Borrie SA, Lansford KL, Barrett TS. Understanding dysrhythmic speech: When rhythm does not matter and learning does not happen. J Acoust Soc Am. 2018 May;143(5):EL379. doi: 10.1121/1.5037620. PMID 29857710
- [Background] Lansford KL, Borrie SA, Barrett TS. Regularity Matters: Unpredictable Speech Degradation Inhibits Adaptation to Dysarthric Speech. J Speech Lang Hear Res. 2019 Nov 20;62(12):4282-4290. doi: 10.1044/2019_JSLHR-19-00055. Print 2019 Dec 18. PMID 31747531
- [Background] Borrie SA, Lansford KL, Barrett TS. Rhythm Perception and Its Role in Perception and Learning of Dysrhythmic Speech. J Speech Lang Hear Res. 2017 Mar 1;60(3):561-570. doi: 10.1044/2016_JSLHR-S-16-0094. PMID 28241307
- [Background] Lansford KL, Borrie SA, Bystricky L. Use of Crowdsourcing to Assess the Ecological Validity of Perceptual-Training Paradigms in Dysarthria. Am J Speech Lang Pathol. 2016 May 1;25(2):233-9. doi: 10.1044/2015_AJSLP-15-0059. PMID 27145295
- [Background] Borrie SA, McAuliffe MJ, Liss JM, Kirk C, O'Beirne GA, Anderson T. Familiarisation conditions and the mechanisms that underlie improved recognition of dysarthric speech. Lang Cogn Process. 2012 Sep 1;27(7-8):1039-1055. doi: 10.1080/01690965.2011.610596. PMID 24009401
- [Background] Borrie SA, Lansford KL, Barrett TS. Generalized Adaptation to Dysarthric Speech. J Speech Lang Hear Res. 2017 Nov 9;60(11):3110-3117. doi: 10.1044/2017_JSLHR-S-17-0127. PMID 29075754
- [Background] Lansford KL, Luhrsen S, Ingvalson EM, Borrie SA. Effects of Familiarization on Intelligibility of Dysarthric Speech in Older Adults With and Without Hearing Loss. Am J Speech Lang Pathol. 2018 Feb 6;27(1):91-98. doi: 10.1044/2017_AJSLP-17-0090. PMID 29305612
- [Background] Hirsch ME, Lansford KL, Barrett TS, Borrie SA. Generalized Learning of Dysarthric Speech Between Male and Female Talkers. J Speech Lang Hear Res. 2021 Feb 17;64(2):444-451. doi: 10.1044/2020_JSLHR-20-00313. Epub 2021 Jan 28. PMID 33508210
- [Background] Lansford KL, Borrie SA, Barrett TS, Flechaus C. When Additional Training Isn't Enough: Further Evidence That Unpredictable Speech Inhibits Adaptation. J Speech Lang Hear Res. 2020 Jun 22;63(6):1700-1711. doi: 10.1044/2020_JSLHR-19-00380. Epub 2020 May 20. PMID 32437259
- [Background] Borrie SA, Lansford KL, Barrett TS. A Clinical Advantage: Experience Informs Recognition and Adaptation to a Novel Talker With Dysarthria. J Speech Lang Hear Res. 2021 May 11;64(5):1503-1514. doi: 10.1044/2021_JSLHR-20-00663. Epub 2021 Apr 8. PMID 33831307
- [Background] Borrie SA, Barrett TS, Yoho SE. Autoscore: An open-source automated tool for scoring listener perception of speech. J Acoust Soc Am. 2019 Jan;145(1):392. doi: 10.1121/1.5087276. PMID 30710955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to COVID-19 limitations at the time of recruitment, initial efforts were focused on recruiting participants 18-50 years. We recruited participants from the Tallahassee, FL and Logan, UT communities. In the later stages of this project, we focused recruitment efforts on older participants aged 55-80 years from the Tallahassee community.
Groups:
- Perceptual Training With Dysarthric Speaker 1: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with dysarthria are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Participants in this condition were assigned to receive perceptual training with a single speaker with ALS (Speaker 1). Pretest/posttest transcription data are used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 2: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with dysarthria are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Participants in this condition were assigned to receive perceptual training with a single speaker with ataxic dysarthria (Speaker 2). Pretest/posttest transcription data are used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 3: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with dysarthria are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Participants in this condition were assigned to receive perceptual training with a single speaker with Parkinson's disease (Speaker 2). Pretest/posttest transcription data are used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 4: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with dysarthria are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Participants in this condition were assigned to receive perceptual training with a single speaker with ALS (Speaker 4). Pretest/posttest transcription data are used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 5: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with dysarthria are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Participants in this condition were assigned to receive perceptual training with a single speaker with PD (Speaker 5). Pretest/posttest transcription data are used to build explanatory models of intelligibility improvement.
Period: Overall Study
Arm/Group | Perceptual Training With Dysarthric Speaker 1 | Perceptual Training With Dysarthric Speaker 2 | Perceptual Training With Dysarthric Speaker 3 | Perceptual Training With Dysarthric Speaker 4 | Perceptual Training With Dysarthric Speaker 5
Started | 49 | 54 | 53 | 32 | 27
Completed | 49 | 54 | 53 | 32 | 27
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Perceptual Training With Dysarthric Speaker 1: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with mixed flaccid-spastic dysarthria due to ALS (Speaker 1) are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 2: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with ataxic dysarthria due to cerebellar degeneration (Speaker 2) are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 3: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with hypokinetic dysarthria due to Parkinson's disease (Speaker 3) are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 4: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with ataxic dysarthria due to cerebellar degeneration (Speaker 4) are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
- Perceptual Training With Dysarthric Speaker 5: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with hypokinetic dysarthria due to Parkinson's disease (Speaker 5) are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
- Total: Total of all reporting groups
Arm/Group | Perceptual Training With Dysarthric Speaker 1 | Perceptual Training With Dysarthric Speaker 2 | Perceptual Training With Dysarthric Speaker 3 | Perceptual Training With Dysarthric Speaker 4 | Perceptual Training With Dysarthric Speaker 5 | Total
Number analyzed (Participants) | 49 | 54 | 53 | 32 | 27 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 54 | 53 | 7 | 2 | 165
  >=65 years | 0 | 0 | 0 | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (7.3) | 22.9 (6.3) | 21.5 (2.9) | 69.28 (4.95) | 70.22 (4.93) | 35 (22)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants did not indicate their sex on intake forms.
  Participants
    Female | 37 | 43 | 43 | 20 | 20 | 163
    Male | 12 | 11 | 10 | 12 | 7 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 12 | 0 | 0 | 30
  Not Hispanic or Latino | 39 | 46 | 41 | 32 | 27 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 3 | 0 | 3 | 11
  White | 44 | 49 | 49 | 32 | 23 | 197
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 3
Working memory [Mean (Standard Deviation); unit: scores on a scale] — We used the NIH Toolbox for all cognitive and sensation measurements. This is an assessment of working memory, in which a participant is asked to recall and sequence different stimuli that are presented visually and via audio. We report participants' age-corrected standard scores are reported. A participant's Age-Corrected Standard score at or near 100 indicates average working memory ability for the age level. Scores around 115 suggest above-average ability. A score of 85 suggests below-average ability. There are no actual minimum or maximum scores.
  scores on a scale | 104 (12) | 104 (10) | 102 (13) | 104 (15) | 109 (17) | 104 (13)
Words-in-Noise [Mean (Standard Deviation); unit: decibels] — We used the Words-in-noise test from the NIH Toolbox, sensation battery. The task requires listeners to identify a series of words presented to each ear individually in a background of increasingly loud noise, thereby reducing the signal-to-noise ratio. The WIN test yields a threshold score for each ear in decibels of signal-to-noise ratio (dB S/N). The best score that can be attained for either ear is -2.0 dB S/N, and the worst score is 26.0 dB S/N. Lower scores are indicative of better performance on this test.
  decibels | 5.6 (1.7) | 5.28 (1.5) | 4.8 (1.1) | 7.9 (4.3) | 8.2 (4.2) | 6.4 (3.3)
Inhibitory control [Mean (Standard Deviation); unit: Scores on a scale] — We used the Flanker inhibitory control measure from the NIH Toolbox website. It is an assessment of inhibitory control and attention. The participant is asked to focus on a particular stimulus while inhibiting attention to the stimuli flanking it. We report participants' age-corrected standard scores are reported. A participant's Age-Corrected Standard score at or near 100 indicates average inhibitory control for the age level. Scores around 115 suggest above-average ability. A score of 85 suggests below-average ability. There are no actual minimum or maximum scores.
  Scores on a scale | 93 (14) | 94 (15) | 90 (17) | 98 (11) | 96 (13) | 94 (15)
Processing speed [Mean (Standard Deviation); unit: Scores on a scale] — We used the Pattern Comparison Processing Speed Test from the NIH Toolbox website to measure processing speed. Participants are asked to quickly determine whether two stimuli are the same or not the same. We report participants' age-corrected standard scores are reported. A participant's Age-Corrected Standard score at or near 100 indicates average processing speed ability for the age level. Scores around 115 suggest above-average ability. A score of 85 suggests below-average ability. There are no actual minimum or maximum scores.
  Scores on a scale | 111 (21) | 115 (19) | 114 (19) | 100 (19) | 100 (20) | 110 (20)
Vocabulary Knowledge [Mean (Standard Deviation); unit: Scores on a scale] — We used the NIH Toolbox picture vocabulary test to measure receptive vocabulary. Participants choose which of four pictures best represents a word presented via audio. We report here the average age-corrected Standard scores based on normative data. A score of 100 indicates vocabulary ability that is average for the age level. Scores around 115 suggest above-average vocabulary ability, while scores around 130 suggest superior ability. Conversely, a score of 85 suggests below-average vocabulary ability. There are no actual minimum or maximum scores.
  Scores on a scale | 105 (14) | 108 (12) | 110 (12) | 112 (10) | 112 (12) | 109 (13)
Cognitive flexibility [Mean (Standard Deviation); unit: Scores on a scale] — We used the dimensional card sort measure of cognitive flexibility from the NIH Toolbox. The participant is asked to match a series of picture pairs to a target picture. We report participants' age-corrected standard scores are reported. A participant's Age-Corrected Standard score at or near 100 indicates average cognitive flexibility ability for the age level. Scores around 115 suggest above-average ability. A score of 85 suggests below-average ability. There are no actual minimum or maximum scores.
  Scores on a scale | 104 (15) | 107 (15) | 104 (17) | 113 (17) | 114 (17) | 107 (16)

OUTCOME MEASURES:

1. Primary Outcome: Pretest Transcription Accuracy
Description: A percentage words correct (PWC) score is tabulated for each listener at pretest. A higher score reflects greater speaker intelligibility (i.e., understanding).
Time Frame: All outcomes were collected during a single data collection session, that lasted no more than 90 minutes. Pretest transcription accuracy is assessed at the pretest, immediately before a single session of perceptual training.
Measure: Mean (Standard Deviation); unit: percentage of words correct
Groups:
- Perceptual Training With Dysarthric Speaker 1; Perceptual Training With Dysarthric Speaker 2; Perceptual Training With Dysarthric Speaker 3; Perceptual Training With Dysarthric Speaker 4; Perceptual Training With Dysarthric Speaker 5: To examine the effect of perceptual training with speakers with dysarthria, we use a standard three-phase perceptual training protocol involving pretest, training, and posttest phases, in which speech samples from a single speaker with dysarthria are utilized for all three phases.
  Perceptual Training: Each listener is familiarized/trained with a single speaker with dysarthria. Pretest/posttest transcription data will be used to build explanatory models of intelligibility improvement.
Arm/Group | Perceptual Training With Dysarthric Speaker 1 | Perceptual Training With Dysarthric Speaker 2 | Perceptual Training With Dysarthric Speaker 3 | Perceptual Training With Dysarthric Speaker 4 | Perceptual Training With Dysarthric Speaker 5
Number analyzed (Participants) | 49 | 54 | 53 | 32 | 27
percentage of words correct | 77.8 (5.4) | 35.3 (7.7) | 52.9 (7.1) | 30 (10.6) | 49.2 (15.4)

2. Primary Outcome: Posttest Transcription Accuracy
Description: A percentage words correct (PWC) score is tabulated for each listener at posttest. Higher scores reflect greater speaker intelligibility (i.e., understanding).
Time Frame: All outcomes were collected during a single data collection session, lasting no longer than 90 minutes. Transcription accuracy at posttest was assessed at posttest, immediately after perceptual training.
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Perceptual Training With Dysarthric Speaker 1 | Perceptual Training With Dysarthric Speaker 2 | Perceptual Training With Dysarthric Speaker 3 | Perceptual Training With Dysarthric Speaker 4 | Perceptual Training With Dysarthric Speaker 5
Number analyzed (Participants) | 49 | 54 | 53 | 32 | 27
percentage of words correct | 84.4 (3.6) | 50 (7.1) | 57.8 (7.8) | 42.2 (12.7) | 51.2 (14.8)

ADVERSE EVENTS:
Time Frame: This is a benign behavioral intervention administered in a single session (day) of 90 minutes.
Arm/Group | Perceptual Training With Dysarthric Speaker 1 | Perceptual Training With Dysarthric Speaker 2 | Perceptual Training With Dysarthric Speaker 3 | Perceptual Training With Dysarthric Speaker 4 | Perceptual Training With Dysarthric Speaker 5
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/54 | 0/53 | 0/32 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/54 | 0/53 | 0/32 | 0/27
Other Adverse Events (participants affected / at risk) | 0/49 | 0/54 | 0/53 | 0/32 | 0/27

LIMITATIONS AND CAVEATS:
While classified as a clinical trial, the aims of this study were to build explanatory models of perceptual learning of dysarthric speech. All participants received perceptual training with one of 5 speakers with dysarthria. The focus of this work was not to establish the efficacy of perceptual training but rather to identify individual listener variables that support perceptual learning. As such, all models were built on individual participant data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT04897711/Prot_SAP_000.pdf